CLINICAL TRIAL: NCT00724932
Title: A Multi-center, Randomized, Parallel-group, Comparative, Active-controlled, Safety-assessor Blinded Trial in Adult Subjects Comparing the Efficacy and Safety of Sugammadex (SCH 900616, ORG 25969) Administered at 1-2 PTC With Neostigmine Administered at Reappearance of T2 in Subjects Undergoing Laparoscopic Cholecystectomy or Appendectomy Under Propofol Anesthesia
Brief Title: Comparison of Sugammadex With Neostigmine During Laparoscopic Cholecystectomy or Appendectomy (P05699)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P05699; 19.4.318 (Other: Organon Protocol ID); MK-8616-002 (Other: Merck Protocol ID); 2007-007951-14 (EudraCT Number)
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Results first posted 2013-04-29 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-04

CONDITIONS: Anesthesia, General
MeSH Terms: interventions — Rocuronium; Sugammadex; Neostigmine; Atropine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugammadex (Experimental): 4.0 mg.kg-1 sugammadex at 1-2 PTC
  Interventions: Drug: Rocuronium; Drug: Sugammadex
- Neostigmine (Experimental): 50 µg.kg-1 neostigmine (with atropine in a ratio of 5:1 for neostigmine:atropine) at reappearance of T2
  Interventions: Drug: Rocuronium; Drug: Neostigmine; Drug: Atropine

INTERVENTIONS:
Drug: Rocuronium — Participants will receive an intravenous (i.v.) single bolus dose of 0.6 mg.kg-1 rocuronium. After this dose, maintenance doses of 0.1-0.2 mg.kg-1 rocuronium may be given.
  Other Names: rocuronium bromide; Esmeron®
Drug: Sugammadex — After the last dose of rocuronium has been administered, participants will receive, according to the randomization, a single bolus dose of 4.0 mg.kg-1 sugammadex at 1-2 PTC.
  Other Names: Org 25969; SCH 900616; MK-8616; Bridion®
  Arms: Sugammadex
Drug: Neostigmine — After the last dose of rocuronium has been administered, participants will receive, according to the randomization, 50 μg.kg-1 neostigmine (with atropine in a ratio of 5:1 for neostigmine:atropine) at reappearance of T2.
  Other Names: Prostigmin®
  Arms: Neostigmine
Drug: Atropine — After the last dose of rocuronium has been administered, participants will receive, according to randomization, 10 μg.kg-1 atropine (with neostigmine in a ratio of 5:1 for neostigmine:atropine) at reappearance of T2.
  Other Names: atropine sulfate
  Arms: Neostigmine

SUMMARY:
The current trial was designed to demonstrate faster recovery from a neuromuscular blockade (NMB) induced by rocuronium after reversal at 1-2 Post Tetanic Count (PTC) by 4.0 mg.kg-1 sugammadex compared to 50 µg.kg-1 neostigmine at reappearance of second twitch (T2) in participants undergoing laparoscopic cholecystectomy or appendectomy under propofol anesthesia, to compare safety and to evaluate operating room and Post Anesthetic Care Unit (PACU) length of stay.

DETAILED DESCRIPTION:
In those surgical procedures where a neuromuscular block is desired for intubation and/or avoid unwanted muscular activity, anesthesiologists may use a more profound NMB until the end of surgery, e.g. in open abdominal procedures or during laparoscopic procedures in order to improve surgical conditions. Reversal with sugammadex at a dose of 4.0 mg.kg-1 at 1-2 PTC after an intubation dose of 0.6 mg.kg-1 or maintenance dosing rocuronium has been found to be both safe and efficacious in previous clinical trials but has never been investigated exclusively in participants undergoing laparoscopic cholecystectomy or appendectomy.

With sugammadex profound muscle relaxation may now be provided right up to the end of the surgical procedure. This may lead to improved Patient Outcomes, such as improvement in the time from end of surgery to the discharge to the PACU. In this multi-center, randomized, parallel-group, active-controlled, safety-assessor blinded trial such benefits will be further investigated.

ELIGIBILITY:
Inclusion Criteria:

* Participants of American Society of Anesthesiologists class 1-3
* Participants of age above or equal to the age of 18 years
* Participants who are scheduled to undergo a laparoscopic cholecystectomy or appendectomy under general anesthesia requiring neuromuscular relaxation with rocuronium, and if applicable, maintenance of neuromuscular blockade
* Participants who have given written informed consent

Exclusion Criteria:

* Participants in whom a difficult intubation because of anatomical malformations is expected
* Participants known or suspected to have neuromuscular disorders affecting NMB
* Participants known or suspected to have a significant renal dysfunction
* Participants known or suspected to have a severe hepatic dysfunction
* Participants known or suspected to have (family) history of malignant hyperthermia
* Participants known or suspected to have an allergy to opioids, muscle relaxants or other medication used during general anesthesia
* Participants in whom the use of neostigmine and/or atropine is contraindicated
* Female participants who are pregnant (pregnancy will be excluded for women both from medical history and by a human chorionic gonadotropin (hCG) test within 24h before surgery, except for women who are not of childbearing potential, i.e. at least 2 years menopausal or have undergone tubal ligation or a hysterectomy)
* Female participants who are breast-feeding
* Participants who participated in another clinical trial not pre-approved by the sponsor, within 30 days of entering into trial 19.4.318 (P05699)
* Participants who have already participated in a sugammadex trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2008-07-16 (Actual); Primary Completion 2009-04-01 (Actual); Study Completion 2009-05-03 (Actual)

REFERENCES:
- [Background] Suresh D, Carter JA, Whitehead JP, Goldhill DR, Flynn PJ. Cardiovascular changes at antagonism of atracurium. Effects of different doses of premixed neostigmine and glycopyrronium in a ratio of 5:1. Anaesthesia. 1991 Oct;46(10):877-80. doi: 10.1111/j.1365-2044.1991.tb09609.x. PMID 1952007
- [Background] Caldwell JE. Reversal of residual neuromuscular block with neostigmine at one to four hours after a single intubating dose of vecuronium. Anesth Analg. 1995 Jun;80(6):1168-74. doi: 10.1097/00000539-199506000-00018. PMID 7762847
- [Background] Irie T, Uekama K. Pharmaceutical applications of cyclodextrins. III. Toxicological issues and safety evaluation. J Pharm Sci. 1997 Feb;86(2):147-62. doi: 10.1021/js960213f. PMID 9040088
- [Background] Apfel CC, Kranke P, Eberhart LH, Roos A, Roewer N. Comparison of predictive models for postoperative nausea and vomiting. Br J Anaesth. 2002 Feb;88(2):234-40. doi: 10.1093/bja/88.2.234. PMID 11883387
- [Background] Apfel CC, Laara E, Koivuranta M, Greim CA, Roewer N. A simplified risk score for predicting postoperative nausea and vomiting: conclusions from cross-validations between two centers. Anesthesiology. 1999 Sep;91(3):693-700. doi: 10.1097/00000542-199909000-00022. PMID 10485781
- [Background] Aldrete JA, Kroulik D. A postanesthetic recovery score. Anesth Analg. 1970 Nov-Dec;49(6):924-34. No abstract available. PMID 5534693
- [Result] Geldner G, Niskanen M, Laurila P, Mizikov V, Hubler M, Beck G, Rietbergen H, Nicolayenko E. A randomised controlled trial comparing sugammadex and neostigmine at different depths of neuromuscular blockade in patients undergoing laparoscopic surgery. Anaesthesia. 2012 Sep;67(9):991-8. doi: 10.1111/j.1365-2044.2012.07197.x. Epub 2012 Jun 14. PMID 22698066

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 10 sites in Germany, Russia, Finland and the United Kingdom between July 2008 and March 2009.
Groups:
- Sugammadex: Participants receiving 4.0 mg.kg-1 sugammadex at 1-2 Post Tetanic Count (PTC)
- Neostigmine: Participants receiving 50 µg.kg-1 neostigmine (with atropine in a ratio of 5:1 for neostigmine: atropine) at reappearance of the second twitch (T2)
Period: Overall Study
Arm/Group | Sugammadex | Neostigmine
Started | 70 | 70
Completed | 65 | 67
Not Completed | 5 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Not treated | 4 | 3

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population consisted of randomized participants who received investigational medicinal product (IMP). Four participants randomized to Sugammadex did not receive IMP and three participants randomized to receive Neostigmine did not receive IMP.
Groups:
- Sugammadex: Participants receiving 4.0 mg.kg-1 sugammadex at 1-2 PTC
- Neostigmine: Participants receiving 50 µg.kg-1 neostigmine (with atropine in a ratio of 5:1 for neostigmine:atropine) at reappearance of T2
- Total: Total of all reporting groups
Arm/Group | Sugammadex | Neostigmine | Total
Number analyzed (Participants) | 66 | 67 | 133
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (16) | 51 (14) | 51 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 43 | 92
  Male | 17 | 24 | 41

OUTCOME MEASURES:

1. Primary Outcome: Time From Start of Administration of Investigational Medicinal Product (IMP, Sugammadex or Neostigmine) to Recovery of the Fourth Twitch/First Twitch (T4/T1) Ratio to 0.9
Description: Neuromuscular functioning was monitored by applying repetitive Train-Of-Four (TOF) electrical stimulations to the ulnar nerve every 15 seconds & assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to the magnitudes (heights) of the first and fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 Ratio (expressed as a decimal of up to 1.0) indicates the extent of recovery from neuromuscular blockade (NMB). In this study, twitch responses were recorded until the T4/T1 Ratio reached >= 0.9, the minimum acceptable ratio that indicated recovery from NMB. A faster time to recovery of the T4/T1 Ratio to 0.9 indicates a faster recovery from NMB.
Time Frame: From start of IMP administration to recovery of T4/T1 ratio to 0.9 (ranging from ~2 minutes to ~9 minutes)
Population: The Intent-To-Treat (ITT) Population consisted of all randomized participants who received IMP and had at least one efficacy measurement. Imputed recovery times were used in cases of missing times.
Measure: Geometric Mean (95% Confidence Interval); unit: minutes
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 66 | 65
minutes | 2.4 [2.1 to 2.7] | 8.4 [7.2 to 9.8]
Statistical Analysis 1: Comparison: Sugammadex vs Neostigmine; To evaluate the efficacy of sugammadex compared to neostigmine, the ratio of the geometric means of time to recovery of the T4/T1 ratio to 0.9 was calculated using a two-way analysis of variance (ANOVA) model adjusted for treatment group and trial site; Test type: Superiority or Other; p < 0.0001, ANOVA — Testing was performed using a two-sided test at the 0.05 significance level. There was only one primary comparison, therefore no adjustment for multiplicity was required; Geometric Mean Ratio (Final Values) = 3.4, 95% CI 2-sided [2.8 to 4.1] — Sugammadex is the numerator and neostigmine the denominator. The estimated value for the geometric mean ratio presents how many times the geometric mean time to recovery of the T4/T1 ratio to 0.9 was faster with sugammadex compared to neostigmine

2. Secondary Outcome: Time From Start of Administration of IMP to Recovery of the T4/T1 Ratio to 0.7
Description: Neuromuscular functioning was monitored by applying repetitive TOF electrical stimulations to the ulnar nerve every 15 seconds & assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to the magnitudes (heights) of the first and fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 Ratio (expressed as a decimal of up to 1.0). A faster time to recovery of the T4/T1 Ratio to 0.7 indicates a faster recovery from NMB.
Time Frame: From start of IMP administration to recovery of T4/T1 Ratio to 0.7 (ranging from ~2 minutes to ~5 minutes)
Population: The ITT Population consisted of all randomized participants who received IMP and had at least one efficacy measurement. Imputed recovery times were used in cases of missing recovery times.
Measure: Geometric Mean (95% Confidence Interval); unit: minutes
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 66 | 65
minutes | 1.6 [1.5 to 1.8] | 4.1 [3.7 to 4.6]
Statistical Analysis 1: Comparison: Sugammadex vs Neostigmine; To evaluate the efficacy of sugammadex compared to neostigmine, the ratio of the geometric means of time to recovery of the T4/T1 ratio to 0.7 was calculated using a two-way ANOVA model adjusted for treatment group and trial site; Test type: Superiority or Other; p < 0.0001, ANOVA — The p-value is not adjusted for multiplicity; Geometric Mean Ratio (Final Values) = 2.5, 95% CI 2-sided [2.1 to 2.8] — Sugammadex is the numerator and neostigmine the denominator. The estimated value for the geometric mean ratio presents how many times the geometric mean time to recovery of the T4/T1 ratio to 0.7 was faster with sugammadex compared to neostigmine

3. Other Pre Specified Outcome: Time From Start of Administration of IMP to Recovery of the T4/T1 Ratio to 0.5 and 0.6
Description: Neuromuscular functioning was monitored by applying repetitive TOF electrical stimulations to the ulnar nerve every 15 seconds & assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to the magnitudes (heights) of the first and fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 Ratio (expressed as a decimal of up to 1.0). Faster times to recovery of the T4/T1 Ratios to 0.5 and 0.6 indicate faster recoveries from NMB.
Time Frame: From start of IMP administration to recovery of T4/T1 Ratio to 0.5 and 0.6 (ranging from ~1 minute to ~4 minutes)
Population: The ITT Population consisted of all randomized participants who received IMP and had at least one efficacy measurement. No imputation was done for missing times to recovery of the T4/T1 ratio to 0.5 and 0.6.
Measure: Geometric Mean (95% Confidence Interval); unit: minutes
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 66 | 65
minutes
  Recovery of T4/T1 Ratio to 0.5 | 1.3 [1.2 to 1.5] | 2.8 [2.5 to 3.1]
  Recovery of T4/T1 Ratio to 0.6 | 1.5 [1.3 to 1.6] | 3.4 [3.1 to 3.8]

4. Other Pre Specified Outcome: Time From Start of Administration of the Last Dose of Rocuronium to Recovery of the T4/T1 Ratio to 0.5, 0.6, 0.7, 0.8 and 0.9
Description: Neuromuscular functioning was monitored by applying repetitive TOF electrical stimulations to the ulnar nerve every 15 seconds & assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to the magnitudes (heights) of the first and fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 Ratio (expressed as a decimal of up to 1.0). A faster time to recovery of the T4/T1 Ratio indicates a faster recovery from NMB.
Time Frame: From start of last dose of rocuronium to recovery of T4/T1 Ratio to 0.5, 0.6, 0.7, 0.8 and 0.9 (ranging from ~12 minutes to ~36 minutes)
Population: The ITT Population consisted of all randomized participants who received IMP and had at least one efficacy measurement. No imputation was done for missing times from administration of last dose of rocuronium to recovery of the T4/T1 ratio to 0.5, 0.6, 0.7, 0.8 and 0.9.
Measure: Geometric Mean (95% Confidence Interval); unit: minutes
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 66 | 65
minutes
  Recovery of T4/T1 ratio to 0.5 | 11.7 [10.1 to 13.6] | 30.0 [26.2 to 34.4]
  Recovery of T4/T1 ratio to 0.6 | 11.9 [10.3 to 13.8] | 30.7 [26.8 to 35.1]
  Recovery of T4/T1 ratio to 0.7 | 12.1 [10.5 to 14.0] | 31.6 [27.7 to 36.0]
  Recovery of T4/T1 ratio to 0.8 | 12.5 [10.8 to 14.3] | 33.2 [29.2 to 37.9]
  Recovery of T4/T1 ratio to 0.9 (N=65, N=61) | 13.3 [11.6 to 15.3] | 35.2 [30.8 to 40.2]

5. Other Pre Specified Outcome: Time From Start of Administration of the Last Dose of Rocuronium to the Time of 1-2 PTC in the 4.0 mg.Kg-1 Sugammadex Group
Description: The time of 1-2 PTC refers to when 1-2 twitches are generated after tetanic stimulation. Time to 1-2 PTC is the time point of the last single twitch >0 or baseline (in case of noise or direct stimulation) within the sequence of a PTC measurement. 1-2 PTC was the target depth of NMB at which sugammadex was to be administered.
Time Frame: From last dose of rocuronium to 1-2 PTC (up to ~9 minutes)
Population: The ITT Population consisted of all randomized participants who received sugammadex and had at least one efficacy measurement. The participants who received neostigmine were not included in this analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: minutes
Groups:
- Sugammadex Only: Participants receiving 4.0 mg.kg-1 sugammadex at 1-2 PTC
Arm/Group | Sugammadex Only
Number analyzed (Participants) | 66
minutes | 8.9 [7.3 to 10.8]

6. Other Pre Specified Outcome: Time From Start of Administration of the Last Dose of Rocuronium to the Time of Reappearance of T2 in the 50 μg.Kg-1 Neostigmine Group
Description: The time of reappearance of T2 refers to when the second twitch reappears after TOF stimulation. Reappearance of T2 was the target depth of NMB at which neostigmine was to be administered.
Time Frame: From last dose of rocuronium to reappearance of T2 (up to ~26 minutes)
Population: The ITT Population consisted of all randomized participants who received neostigmine and had at least one efficacy measurement. The participants who received sugammadex were not included in this analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: minutes
Groups:
- Neostigmine Only: Participants receiving 50 µg.kg-1 neostigmine (with atropine in a ratio of 5:1 for neostigmine:atropine) at reappearance of T2
Arm/Group | Neostigmine Only
Number analyzed (Participants) | 65
minutes | 25.6 [21.8 to 30.0]

7. Other Pre Specified Outcome: Mean Systolic Blood Pressure
Description: Systolic Blood Pressure was measured at screening, before start of rocuronium administration, before start of IMP administration, at 2, 5, 10, 30 minutes post-IMP administration, and at the post-anesthetic visit (the day after surgery).
Time Frame: At screening, pre-rocuronium, pre-IMP, at 2, 5, 10, and 30 minutes post-IMP, and at the post-anesthetic visit (the day after surgery)
Population: The AST Population consisted of all randomized participants who received IMP.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 66 | 67
mm Hg
  Screening | 132.7 (17.7) | 133.9 (19.1)
  Pre-rocuronium | 98.2 (13.9) | 101.6 (18.2)
  Pre-IMP | 122.1 (16.5) | 121.3 (18.8)
  2 minutes post-IMP (N=65, N=65) | 122.5 (18.8) | 122.5 (20.4)
  5 minutes post-IMP | 122.6 (17.7) | 118.0 (22.3)
  10 minutes post-IMP (N=66, N=66) | 124.0 (17.8) | 119.3 (23.7)
  30 minutes post-IMP (N=65, N=66) | 132.9 (17.4) | 131.7 (23.0)
  Post-anesthetic visit (N=66, N=66) | 127.3 (16.6) | 125.4 (17.1)

8. Other Pre Specified Outcome: Mean Diastolic Blood Pressure
Description: Diastolic Blood Pressure was measured at screening, before start of rocuronium administration, before start of IMP administration, at 2, 5, 10, 30 minutes post-IMP administration, and at the post-anesthetic visit (the day after surgery).
Time Frame: as for outcome 7
Population: The AST Population consisted of all randomized participants who received IMP.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 66 | 67
mm Hg
  Screening | 80.9 (9.9) | 82.8 (9.4)
  Pre-rocuronium | 58.2 (11.6) | 58.3 (10.1)
  Pre-IMP | 72.8 (12.1) | 72.5 (12.8)
  2 minutes post-IMP (N=65, N=65) | 73.4 (11.8) | 72.6 (11.8)
  5 minutes post-IMP | 72.4 (11.4) | 69.2 (13.5)
  10 minutes post-IMP (N=66, N=66) | 71.8 (12.8) | 68.7 (14.9)
  30 minutes post-IMP (N=65, N=66) | 74.3 (10.9) | 73.1 (13.5)
  Post-anesthetic visit (N=66, N=66) | 76.7 (9.4) | 75.2 (10.8)

9. Other Pre Specified Outcome: Mean Heart Rate
Description: Heart Rate was measured at screening, before start of rocuronium administration, before start of IMP administration, at 2, 5, 10, 30 minutes post-IMP administration, and at the post-anesthetic visit (the day after surgery).
Time Frame: as for outcome 7
Population: The AST Population consisted of all randomized participants who received IMP.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 66 | 67
beats per minute
  Screening | 72.9 (11.0) | 74.6 (11.4)
  Pre-rocuronium | 63.4 (13.4) | 63.6 (12.4)
  Pre-IMP | 68.3 (11.0) | 68.0 (12.3)
  2 minutes post-IMP (N=65, N=65) | 66.0 (12.4) | 65.3 (12.4)
  5 minutes post-IMP | 64.9 (12.3) | 57.1 (10.8)
  10 minutes post-IMP (N=66, N=66) | 67.3 (12.4) | 56.3 (11.4)
  30 minutes post-IMP (N=65, N=66) | 73.1 (12.2) | 65.1 (11.2)
  Post-anesthetic visit (N=66, N=66) | 72.7 (11.7) | 71.9 (71.9)

10. Secondary Outcome: Time From Start of Administration of IMP to Recovery of the T4/T1 Ratio to 0.8
Description: Neuromuscular functioning was monitored by applying repetitive TOF electrical stimulations to the ulnar nerve every 15 seconds & assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to the magnitudes (heights) of the first and fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 Ratio (expressed as a decimal of up to 1.0). A faster time to recovery of the T4/T1 Ratio to 0.8 indicates a faster recovery from NMB.
Time Frame: From start of IMP administration to recovery of T4/T1 Ratio to 0.8 (ranging from ~2 minutes to ~6 minutes)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: minutes
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 66 | 65
minutes | 1.9 [1.7 to 2.1] | 5.6 [4.9 to 6.3]
Statistical Analysis 1: Comparison: Sugammadex vs Neostigmine; To evaluate the efficacy of sugammadex compared to neostigmine, the ratio of the geometric means of time to recovery of the T4/T1 ratio to 0.8 was calculated using a two-way ANOVA model adjusted for treatment group and trial site; Test type: Superiority or Other; p < 0.0001, ANOVA — The p-value is not adjusted for multiplicity; Geometric Mean Ratio (Final Values) = 2.9, 95% CI 2-sided [2.5 to 3.4] — Sugammadex is the numerator and neostigmine the denominator. The estimated value for the geometric mean ratio presents how many times the geometric mean time to recovery of the T4/T1 ratio to 0.8 was faster with sugammadex compared to neostigmine

11. Other Pre Specified Outcome: Number of Participants Who Had Physical Examinations
Description: Physical examinations were to be conducted at screening (within 7 days prior to surgery) and at the post-anesthetic visit (the day after surgery).
Time Frame: At screening (within 7 days prior to surgery) and at the post-anesthetic visit (the day after surgery)
Population: The AST Population consisted of all randomized participants who received IMP. As there was no specific physical examination case report form used in this study, data on whether or not a physical examination was conducted were not recorded.
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 0 | 0

12. Other Pre Specified Outcome: Number of Participants With Train-of-Four- (TOF-) Watch® SX and Arm Board Related Adverse Events
Description: Events were to be collected for the entire period of neuromuscular transmission monitoring and were defined as an occurrence that resulted or could have resulted in: death; a serious deterioration in the state of health of a user; an occurrence which might, if it recurred, lead to death or serious deterioration in health; inaccuracy as well as any inadequacy in the labeling or instructions which could cause misuse or incorrect maintenance or adjustment which might lead to a death or serious deterioration in health; an examination of the medical device or the information supplied with the medical device indicated some factor with the potential for an incident involving death or serious deterioration in health; malfunction or deterioration in characteristics and/or performance of a medical device, which might lead to death, or serious deterioration in health; technical/medical recalls involving risk of death or serious deterioration in the state of health of the user.
Time Frame: From induction of anesthesia to recovery from NMB (up to ~3 hours)
Population: The AST Population consisted of all randomized participants who received IMP.
Measure: Number; unit: participants
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 66 | 67
participants | 0 | 0

13. Other Pre Specified Outcome: Number of Participants With Reoccurrence of Neuromuscular Blockade Based on the Train-of-Four- (TOF-) Watch® SX Recording (i.e. a Decline in T4/T1 Ratio From >=0.9 to <0.8 in at Least Three Consecutive TOF Values)
Description: Neuromuscular functioning was monitored by applying repetitive TOF electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to the magnitudes (heights) of the 1st and 4th twitches, respectively, after TOF stimulation. The T4/T1 Ratio is expressed as a decimal of up to 1.0. A higher ratio indicates greater recovery from NMB. A decline in the T4/T1 ratio from >=0.9 (indicating a recovery from NMB) to <0.8 for at least three consecutive TOF values was considered to be a reoccurrence of NMB.
Time Frame: Up to 30 minutes after IMP administration
Population: The ITT Population consisted of all randomized participants who received IMP and had at least one efficacy measurement.
Measure: Number; unit: participants
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 66 | 65
participants | 0 | 0

14. Other Pre Specified Outcome: Number of Participants With Clinical Evidence of Reoccurrence of Neuromuscular Blockade or Residual Neuromuscular Blockade (Routine Oxygen Saturation by Pulse Oximetry and Breath Frequency Measurement)
Description: Clinical evidence of reoccurrence of NMB or residual NMB was assessed by oxygen saturation (by pulse oximetry) and breath frequency measurements as per routine practice after anesthesia and neuromuscular monitoring.
Time Frame: Up to 24 hours after IMP administration
Population: The AST Population consisted of all randomized participants who received IMP.
Measure: Number; unit: participants
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 66 | 67
participants | 1 | 0

15. Other Pre Specified Outcome: Number of Participants With Events Due to a Possible Interaction of Sugammadex With Endogenous Compounds or With Exogenous Compounds Other Than Rocuronium
Description: Any evidence of events due to a possible interaction of sugammadex with endogenous compounds or with exogenous compounds other than rocuronium, was to be recorded.
Time Frame: Up to 7 days after IMP administration
Population: The AST Population consisted of all randomized participants who received sugammadex. Participants who received neostigmine were excluded from this analysis.
Measure: Number; unit: participants
Arm/Group | Sugammadex Only
Number analyzed (Participants) | 66
participants | 0

16. Other Pre Specified Outcome: Monitoring of Clinical Signs of Recovery According to Routine Anesthetic Procedures at the Trial Sites
Description: The monitoring of clinical signs of recovery was to be conducted based on the routine anesthetic procedures at each site.
Time Frame: Up to PACU discharge (up to ~4.5 hours)
Population: The AST Population consisted of all randomized participants who received IMP.
Measure: Number; unit: participants
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 66 | 67
participants | NA — This was a site-specific outcome measure. Data were collected at each site, but were not collected on a case report form and were not analyzed. | NA — This was a site-specific outcome measure. Data were collected at each site, but were not collected on a case report form and were not analyzed.

17. Other Pre Specified Outcome: Number of Female Participants or Partners of Male Participants Who Became Pregnant During Study
Description: Thirty days after administration of IMP, female participants of childbearing potential were asked whether they became pregnant during the trial and male participants were asked whether their partner (if of childbearing potential) became pregnant during the trial.
Time Frame: Up to 30 days after IMP administration
Population: The AST Population consisted of all randomized participants who received IMP.
Measure: Number; unit: participants
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 66 | 67
participants | 0 | 0

18. Other Pre Specified Outcome: Time From Operating Room Admission to Operating Room Discharge Ready
Description: The time of Operating Room admission was defined as the time at which the participant was physically placed into the Operating Room. The time of Operating Room discharge ready was defined as time at which the participant had T4/T1 ratio of ≥0.9 and the participant's wound dressing was in place.
Time Frame: From Operating Room admission to Operating Room discharge ready (up to ~3 hours)
Population: The ITT Population consisted of all randomized participants who received IMP and had at least one efficacy measurement.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 66 | 65
minutes | 154 (46) [137 to 159] | 165 (55) [144 to 170]

19. Other Pre Specified Outcome: Time From Operating Room Admission to Actual Operating Room Discharge
Description: The time of Operating Room admission was defined as the time at which the participant was physically placed into the Operating Room. The time of Operating Room discharge was defined as the actual time the participant was discharged from the Operating Room.
Time Frame: From Operating Room admission to actual Operating Room discharge (up to ~3 hours)
Population: The ITT Population consisted of all randomized participants who received IMP and had at least one efficacy measurement.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 66 | 64
minutes | 158 (47) | 169 (58)

20. Other Pre Specified Outcome: Time From Operating Room Discharge Ready to Actual Operating Room Discharge
Description: The time of Operating Room discharge ready was defined as time at which the participant had T4/T1 ratio of >=0.9 and the participant's wound dressing was in place. The time of Operating Room discharge was defined as the actual time the participant was discharged from the Operating Room.
Time Frame: From Operating Room discharge ready to actual Operating Room discharge (up to ~5 minutes)
Population: The ITT Population consisted of all randomized participants who received IMP and had at least one efficacy measurement.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 66 | 64
minutes | 4 (5) | 5 (6)

21. Other Pre Specified Outcome: Time From Start of IMP Administration to T4/T1 Ratio of <=0.60, >0.60 - <=0.70, >0.70 - <=0.80, >0.80 - <0.90 and >=0.90
Description: The time of IMP administration was defined as the actual time at which IMP administration was started.
Time Frame: From start of IMP administration to recovery of the T4/T1 ratio to the designated value (ranging from ~1 minute to ~10 minutes)
Population: The ITT Population consisted of all randomized participants who received IMP and had at least one efficacy measurement. Data not collected. In Protocol Amendment 2, this outcome measure was removed.
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 0 | 0

22. Other Pre Specified Outcome: Time From Start of IMP Administration to Tracheal Extubation
Description: The time of IMP administration was defined as the actual time at which IMP administration was started. The time of tracheal extubation was defined as the actual time at which the participant was extubated.
Time Frame: From start of IMP administration to tracheal extubation (up to ~21 minutes)
Population: The ITT Population consisted of all randomized participants who received IMP and had at least one efficacy measurement.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 66 | 65
minutes | 14 (8) | 21 (11)

23. Other Pre Specified Outcome: Time From Start of IMP Administration to Operating Room Discharge Ready
Description: The time of IMP administration was defined as the actual time at which IMP administration was started. The time of Operating Room discharge ready was defined as time at which the participant had T4/T1 ratio of >=0.9 and the participant's wound dressing was in place.
Time Frame: From start of IMP administration to Operating Room discharge ready (up to ~21 minutes)
Population: The ITT Population consisted of all randomized participants who received IMP and had at least one efficacy measurement.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 66 | 65
minutes | 15 (8) | 21 (11)

24. Other Pre Specified Outcome: Time From Start of IMP Administration to Actual Operating Room Discharge
Description: The time of IMP administration was defined as the actual time at which IMP administration was started. The time of Operating Room discharge was defined as the actual time at which the participant was discharged from the Operating Room.
Time Frame: From start of IMP administration to actual Operating Room discharge (up to ~26 minutes)
Population: The ITT Population consisted of all randomized participants who received IMP and had at least one efficacy measurement.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 66 | 64
minutes | 19 (9) | 26 (13)

25. Other Pre Specified Outcome: Time From Tracheal Extubation to Operating Room Discharge Ready
Description: The time of tracheal extubation was defined as the actual time at which the participant was extubated. The time of Operating Room discharge ready was defined as time at which the participant had T4/T1 ratio of >=0.9 and the participant's wound dressing was in place.
Time Frame: From tracheal extubation to Operating Room discharge ready (up to ~1 minute)
Population: The ITT Population consisted of all randomized participants who received IMP and had at least one efficacy measurement.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 66 | 65
minutes | 1 (6) | 0 (6)

26. Other Pre Specified Outcome: Time From Tracheal Extubation to Actual Operating Room Discharge
Description: The time of tracheal extubation was defined as the actual time at which the participant was extubated. The time of Operating Room discharge was defined as the actual time at which the participant was discharged from the Operating Room.
Time Frame: From tracheal extubation to actual OR discharge (up to ~5 minutes)
Population: The ITT Population consisted of all randomized participants who received IMP and had at least one efficacy measurement.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 66 | 64
minutes | 5 (7) | 5 (6)

27. Other Pre Specified Outcome: Time From Operating Room Discharge Ready to Post Anesthetic Care Unit (PACU) Discharge Ready
Description: The time of Operating Room discharge ready was defined as time at which the participant had T4/T1 ratio of >=0.9 and the participant's wound dressing was in place. The time of PACU discharge ready was defined as the time at which the participant had a Modified Aldrete Score >=9. The Modified Aldrete Score was to be assessed at PACU arrival, at 5, 15, 30, 45, 60 minutes after PACU arrival and every 15 minutes thereafter (if applicable) until the participant was ready to be discharged from the PACU. The Modified Aldrete Postoperative Recovery Score (range = 0-10) is calculated based on scores of 0 to 2 each for Activity, Respiration, Circulation, Consciousness and Oxygen Saturation, with a higher score indicating increased postoperative recovery.
Time Frame: From Operating Room discharge ready to PACU discharge ready (up to ~33 minutes)
Population: The ITT Population consisted of all randomized participants who received IMP and had at least one efficacy measurement.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 66 | 65
minutes | 28 (27) | 33 (40)

28. Other Pre Specified Outcome: Time From Operating Room Discharge Ready to Actual PACU Discharge
Description: The time of Operating Room discharge ready was defined as time at which the participant had T4/T1 ratio of >=0.9 and the participant's wound dressing was in place. The time of PACU discharge was defined as the actual time the participant was discharged from the PACU.
Time Frame: From Operating Room discharge ready to actual PACU discharge (up to ~4.5 hours)
Population: The ITT Population consisted of all randomized participants who received IMP and had at least one efficacy measurement.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 66 | 65
minutes | 268 (348) | 210 (283)

29. Other Pre Specified Outcome: Time From Actual Operating Room Discharge to PACU Discharge Ready
Description: The time of Operating Room discharge was defined as the actual time the participant was discharged from the Operating Room. The time of PACU discharge ready was defined as the time at which the participant had a Modified Aldrete Score >=9. The Modified Aldrete Score was to be assessed at PACU arrival, at 5, 15, 30, 45, 60 minutes after PACU arrival and every 15 minutes thereafter (if applicable) until the participant was ready to be discharged from the PACU. The Modified Aldrete Postoperative Recovery Score (range = 0-10) is calculated based on scores of 0 to 2 each for Activity, Respiration, Circulation, Consciousness and Oxygen Saturation, with a higher score indicating increased postoperative recovery.
Time Frame: From actual Operating Room discharge to PACU discharge ready (up to ~30 minutes)
Population: The ITT Population consisted of all randomized participants who received IMP and had at least one efficacy measurement.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 66 | 64
minutes | 24 (28) | 29 (40)

30. Other Pre Specified Outcome: Time From Actual Operating Room Discharge to Actual PACU Discharge
Description: The time of Operating Room discharge was defined as the actual time the participant was discharged from the Operating Room. The time of PACU discharge was defined as the actual time the participant was discharged from the PACU.
Time Frame: From actual Operating Room discharge to actual PACU discharge (up to ~4.4 hours)
Population: The ITT Population consisted of all randomized participants who received IMP and had at least one efficacy measurement.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 66 | 64
minutes | 264 (347) | 207 (284)

31. Other Pre Specified Outcome: Time From PACU Admit to PACU Discharge Ready
Description: The time of PACU admit was defined as the actual time the participant was admitted to the PACU. The time of PACU discharge ready was defined as the time at which the participant had a Modified Aldrete Score >=9. The Modified Aldrete Score was to be assessed at PACU arrival, at 5, 15, 30, 45, 60 minutes after PACU arrival and every 15 minutes thereafter (if applicable) until the participant was ready to be discharged from the PACU. The Modified Aldrete Postoperative Recovery Score (range = 0-10) is calculated based on scores of 0 to 2 each for Activity, Respiration, Circulation, Consciousness and Oxygen Saturation, with a higher score indicating increased postoperative recovery.
Time Frame: From PACU admit to PACU discharge ready (up to ~25 minutes)
Population: The ITT Population consisted of all randomized participants who received IMP and had at least one efficacy measurement.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 66 | 64
minutes | 20 (28) | 25 (40)

32. Other Pre Specified Outcome: Time From PACU Admit to Actual PACU Discharge
Description: The time of PACU admit was defined as the actual time the participant was admitted to the PACU. The time of PACU discharge was defined as the actual time the participant was discharged from the PACU.
Time Frame: From PACU admit to actual PACU discharge (up to ~4.3 hours)
Population: The ITT Population consisted of all randomized participants who received IMP and had at least one efficacy measurement.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 66 | 64
minutes | 260 (347) | 203 (284)

33. Secondary Outcome: Number of Participants Who Experienced Pre-treatment Serious Adverse Events (SAEs) and Post-treatment SAEs
Description: An SAE is defined as any untoward medical occurrence that at any dose: results in death; is life-threatening; requires in-patient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; or is a congenital anomaly/birth defect.
  Participants were monitored for occurrence SAEs for up to 7 days after last dose IMP. Pre-treatment refers to the period from signing of the informed consent up to start of IMP administration. Post-treatment refers to the period from start of IMP administration to 7 days after IMP administration.
Time Frame: From signing of informed consent to end of trial (7 days after surgery)
Population: The All-Subjects-Treated (AST) Population consisted of all randomized participants who received IMP.
Measure: Number; unit: participants
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 66 | 67
participants
  Pre-treatment SAE | 1 | 0
  Post-treatment SAE | 4 | 6

34. Secondary Outcome: Number of Participants Who Experienced Pre-treatment Non-serious Adverse Events (AEs) and Post-treatment Non-serious AEs
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body, whether or not considered related to the use of the product. Participants were monitored for occurrence AEs for up to 7 days after last dose IMP. Pre-treatment refers to the period from signing of the informed consent up to start of IMP administration. Post-treatment refers to the period from start of IMP administration to 7 days after IMP administration.
Time Frame: From signing of informed consent to end of trial (7 days after surgery)
Population: The AST Population consisted of all randomized participants who received IMP.
Measure: Number; unit: participants
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 66 | 67
participants
  Pre-treatment non-serious AE | 38 | 34
  Post-treatment non-serious AE | 65 | 65

ADVERSE EVENTS:
Time Frame: Up to 7 days after IMP administration
Description: The AST Population consisted of all randomized participants who received IMP.
  * Serious Adverse Events (SAEs) include both pre-treatment (from signing of informed consent to start of IMP administration) and post-treatment (from start of IMP administration to 7 days after IMP administration) SAEs.
Groups:
- Neostigmine: Participants receiving 50 µg.kg-1 neostigmine (with atropine in a ratio of 5:1 for neostigmine: atropine) at reappearance of T2
Arm/Group | Sugammadex | Neostigmine
Serious Adverse Events (participants affected / at risk) | 5/66 | 6/67
Other Adverse Events (participants affected / at risk) | 64/66 | 63/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex (N=66) | Neostigmine (N=67)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Operative haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural vomiting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sedation (Nervous system disorders) | 0 (0) | 1 (1)
Vascular calcification (Vascular disorders) | 1 (1) | 0 (0)
Vascular thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex (N=66) | Neostigmine (N=67)
Abdominal Pain (Gastrointestinal disorders) | 5 (5) | 4 (4)
Constipation (Gastrointestinal disorders) | 6 (6) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 4 (4)
Flatulence (Gastrointestinal disorders) | 2 (2) | 4 (4)
Nausea (Gastrointestinal disorders) | 16 (17) | 12 (13)
Vomiting (Gastrointestinal disorders) | 8 (8) | 7 (7)
Anaesthetic complication cardiac (Injury, poisoning and procedural complications) | 1 (1) | 9 (9)
Procedural nausea (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
Procedural pain (Injury, poisoning and procedural complications) | 60 (70) | 60 (72)
Procedural vomiting (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
C-reactive protein increased (Investigations) | 8 (8) | 6 (6)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No